CLINICAL TRIAL: NCT05762211
Title: A Multi-center Randomized, Double Blinded Phase IIb Trial Evaluating Oral Pooled Fecal Microbiotherapy MaaT033 to Prevent Allogeneic Hematopoietic Cell Transplantation Complications (PHOEBUS Trial)
Brief Title: Oral Pooled Fecal Microbiotherapy to Prevent Allogeneic Hematopoietic Cell Transplantation Complications (PHOEBUS Trial)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MaaT Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MPOH08
Record Dates: First submitted 2023-01-27; First posted 2023-03-09 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Transplant Complication

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral pooled fecal microbiotherapy - MaaT033 (Experimental): 3 capsules per day
  Interventions: Drug: Pooled allogeneic fecal microbiotherapy
- Placebo capsule (Placebo Comparator): 3 capsules per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pooled allogeneic fecal microbiotherapy — Capsule for oral use
  Other Names: MaaT033
  Arms: Oral pooled fecal microbiotherapy - MaaT033
Drug: Placebo — Capsule for oral use
  Arms: Placebo capsule

SUMMARY:
This randomized, placebo-controlled phase IIb study (PHOEBUS trial) aims to evaluate the activity of fecal microbiotherapy MaaT033 to improve survival through the prevention of transplant-related complications in eligible alloHCT patients

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years old
* Presence of a hematologic malignancy for which an alloHCT is indicated with a reduced toxicity or reduced intensity conditioning regimen
* Patients with polynuclear neutrophils > 0.5 G/L
* Patients having received wide spectrum antibiotics within the last 90 days prior to inclusion
* Karnofsky index ≥ 70%
* Availability of a sibling donor, an unrelated stem-cell donor or a familial haploidentical donor
* Written informed consent

Exclusion Criteria:

* Patients planned to receive a non-myeloablative conditioning regimen (2 Gray total body irradiation (TBI) +/- purine analog, fludarabine + cyclophosphamide or equivalent)
* Patients planned to receive a conventional myeloablative conditioning regimen (e.g. high dose cyclophosphamide and high dose TBI (≥10Gy); high dose busulfan (12.8 mg/kg IV) + high dose cyclophosphamide)
* Patients receiving a manipulated graft (in-vitro T-cell depletion)
* Patients planned to receive a conditioning regimen with alemtuzumab
* Patients planned to receive alloHCT with cord blood cells
* Patients planned to receive alloHCT from unrelated donor with >= 3/10 HLA-mismatches
* Patients receiving a large spectrum antibiotic at time of randomization
* Patients planned to receive vedolizumab or abatacept for GvHD prophylaxis
* Creatinine clearance <30 mL/min
* Bilirubin or amino-transferases abnormalities contra-indicating alloHCT
* Cardiac ejection fraction less than 40%
* Pulmonary impairment with <50% lung carbon monoxide diffusing capacity (DLCO)
* Pregnancy
* Confirmed or suspected intestinal ischemia
* Confirmed or suspected toxic megacolon or gastrointestinal perforation
* Any history of gastro-intestinal surgery in the past 3 months
* Any history of chronic digestive disease (Crohn's disease, ulcerative colitis, inflammatory bowel disease or other relevant digestive condition according to physician's judgement)
* Known allergy or intolerance to trehalose or maltodextrin
* Patients with EBV-IgG negative serology
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the subject; or interfere with interpretation of study data.
* Vulnerable patients such as: persons deprived of liberty, persons in Intensive Care Unit unable to provide informed consent prior to the intervention.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 12 months post alloHCT
  To compare the efficacy of MaaT033 with its placebo on OS at 12 months after alloHCT

SECONDARY OUTCOMES:
Restoration of gut microbiota diversity | 12 months post alloHCT
  To evaluate MaaT033 efficacy in gut microbiota diversity restoration using alpha-diversity (Richness index)
grade 2-4 acute GvHD | 6 months post alloHCT
  To evaluate the cumulative incidence of grade 2-4 acute GvHD within 6 months after alloHCT
grade 3-4 acute GvHD | 12 months post alloHCT
  To evaluate the cumulative incidence of grade 3-4 severe acute GvHD within 12+
  + months after alloHCT
Non-relapse mortality | 12 months post alloHCT
  To evaluate the cumulative incidence of non-relapse mortality within 12 months after alloHCT
Infectious-related mortality | 12 months post alloHCT
  To evaluate the cumulative incidence of infectious-related mortality within 12 months after alloHCT
GvHD-related mortality | 12 months post alloHCT
  To evaluate the cumulative incidence of GvHD-related mortality within 12 months after alloHCT
GRFS | 12 months post alloHCT
  To evaluate GvHD-free relapse-free survival (GRFS) at 12 months after alloHCT
Quality of life questionnaire | 12 months post alloHCT
  To evaluate the Quality of Life (EORTC QLQ C30 questionnaire)
Quality of life questionnaire | 12 months post alloHCT
  To evaluate the Quality of Life (FACT-BMT questionnaire)
Proportion of patients with severe infections | 6 months after alloHCT
  To evaluate the proportion of patients with severe infections defined by NCI-CTCAE ≥ Grade 3 within 6 months after alloHCT
Proportion of patients who have discontinued immune suppression therapies | 12 months after alloHCT
  To evaluate the proportion of patients who have discontinued immune suppression therapies including standard of care GvHD prophylaxis and steroid treatment
Time to platelet engraftment | 12 months after alloHCT
  Time to the first of 3 consecutive days of absolute neutrophil counts ≥ 0.5 G/L after alloHCT
Time to neutrophil engraftment | 12 months after alloHCT
  Time to the first of 3 consecutive days of platelet counts ≥ 20 G/L after alloHCT
Safety: incidence of AEs | 12 months after alloHCT
  To evaluate MaaT033 safety

CONTACTS AND LOCATIONS:
Overall Officials: Florent Malard, MD, PhD, Principal Investigator — APHP
Locations (54):
- Belgium (7):
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - AZ Sint - Jan Brugge, Bruges
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Cliniques Universitaires Saint-Luc, Leuven
  - Algemeen Ziekenhuis Delta - Campus Rumbeke, Roeselare
- France (20):
  - CHU Angers, Angers
  - CHU Besançon, Besançon
  - CHU Caen, Caen
  - CHU Grenoble, La Tronche
  - CHRU Lille, Lille
  - Centre Hospitalier Universitaire Limoges, Limoges
  - Institut Paoli Calmettes, Marseille
  - Hôpital Saint-Eloi, Montpellier
  - CHU Nantes Hôtel Dieu, Nantes
  - Hôpital l'Archet, Nice
  - Hôpital Saint-Louis, Paris
  - Hôpital St Antoine, Paris
  - Hôpital Haut-Lévêque, Pessac
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - CHU Rennes - Hôpital Pontchaillou, Rennes
  - CHU St Etienne, Saint-Priest-en-Jarez
  - IUCT Toulouse, Toulouse
  - Centre Hospitalier Régional Universitaire de Tours, Tours
  - CHU Tours, Tours
- Germany (11):
  - Universitätsklinikum Augsburg, Augsburg
  - Helios Klinikum Berlin-Buch, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum des Saarlandes, Hombourg
  - Universitätsklinikum Schleswig-Holstein - Campus Kiel, Kiel
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsmedizin Mannheim, Mannheim
  - Klinikum rechts der Isar der Technischen Universität, München
  - Universitätsklinikum Ulm, Ulm
- Universitair Medisch Centrum Groningen, Groningen, Netherlands
- Spain (14):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Institut Català d'Oncologia - Hospital Duran i Reynals (ICO L'Hospitalet), Barcelona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda
  - Hospital General Universitario Morales Meseguer, Murcia
  - Clinica Universidad de Navarra - Pamplona, Pamplona
  - Complejo Asistencial Universitario de Salamanca - Hospital Clínico, Salamanca
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Clínico Universitario de Valencia Avenida Blasco Ibáñez, Valencia
  - Hospital Universitario La Fe, Valencia
- Cardiff and Vale University Health Board, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No